CLINICAL TRIAL: NCT00219310
Title: A Study to Determine the Safety and Efficacy of Famciclovir in the Episodic and Suppressive Treatment of Recurrent Genital Herpes (RGH). The Study Will Also Evaluate Quality of Life and Patient Satisfaction
Brief Title: RELIEF: Randomized Episodic Versus Long-Term Suppression Experience With Famciclovir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFAM810AUS07
Record Dates: First submitted 2005-09-21; First posted 2005-09-22 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Recurrent Genital Herpes (RGH)
Keywords: Recurrent Genital Herpes (RGH), famciclovir, episodic treatment, suppressive treatment, Polymerase Chain Reaction (PCR).
MeSH Terms: conditions — Herpes Genitalis; Pathologic Complete Response | interventions — Famciclovir

INTERVENTIONS:
Drug: Famciclovir

SUMMARY:
This trial will assess whether RGH patients who have two recurrent episodes within a three month period would benefit from suppressive treatment and whether patients prefer episodic therapy or suppressive therapy for the treatment of their RGH.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are immunocompetent and who have had 4 or more episodes of Recurrent Genital Herpes (RGH) in the last 12 months.

  * Patients with active HSV-2 or HSV-1 infection as confirmed by Polymerase Chain Reaction (PCR).
  * Patients with active symptoms (i.e., itching, burning, tingling, aching, tenderness, rash or pain) associated with a recurrent episode of genital herpes

Exclusion Criteria:

* • Female patients who are pregnant or breast-feeding.

  * Current, history or suspicion of liver disease or kidney disease.
  * HIV infected (as confirmed by positive HIV serology).

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Time (days from randomizations) to first recurrence of symptoms of recurrent genital herpes confirmed by PCR.

SECONDARY OUTCOMES:
Change in total score of the Recurrent Genital Herpes Quality of Life.
Safety assessed by adverse events.
Time to first recurrence of genital herpes.
Number of genital herpes recurrences confirmed by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Bartlett BL, Tyring SK, Fife K, Gnann JW Jr, Hadala JT, Kianifard F, Berber E. Famciclovir treatment options for patients with frequent outbreaks of recurrent genital herpes: the RELIEF trial. J Clin Virol. 2008 Oct;43(2):190-5. doi: 10.1016/j.jcv.2008.06.004. Epub 2008 Jul 14. PMID 18621575